CLINICAL TRIAL: NCT04973800
Title: The Effect of 28-day Simvastatin Administration on Emotional Processing, Reward Learning, Working Memory, and Salivary Cortisol in Healthy Volunteers At-risk for Depression
Brief Title: Simvastatin and Emotional Processing (OxSTEP)
Acronym: OxSTEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R73946/RE001
Record Dates: First submitted 2021-06-28; First posted 2021-07-22 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2022-08

CONDITIONS: Depression; Inflammation
MeSH Terms: conditions — Depression; Inflammation | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The simvastatin and the placebo tablets will be sourced from the Oxford Pharmacy Stores and HSC (www.hsconline.co.uk) respectively, and will be encapsulated at the Neurosciences Building according to our standard operating procedure (APPENDIX D: Neurosciences, SOP Number: Encapsulation Version 2: 22.10.2012). Blinding will be achieved by the identical matching of the simvastatin and placebo treatments. Participants will not be aware of the treatment that they will be receiving; neither will the researchers, as this study is double-blind. Allocation of treatments will be recorded on a randomisation list, which will be updated when each new participant enters the randomised phase. The list will be held at the Neurosciences Building by a scientist uninvolved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm: Simvastatin (Experimental): Simvastatin 20mg ON PO for 28-30 days
  Interventions: Drug: Simvastatin 20mg
- Control arm: Placebo (Placebo Comparator): Sucrose placebo ON PO for 28-30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin 20mg — Simvastatin 20mg ON PO for 28-30 days
  Arms: Experimental arm: Simvastatin
Drug: Placebo — Sucrose placebo ON PO for 28-30 days
  Arms: Control arm: Placebo

SUMMARY:
Simvastatin is being employed because it is a 'statin'. As a drug class, statins have broad anti-inflammatory properties. Low-level inflammation is thought to be a potentially important mediator of the effects of psychosocial stress (including loneliness) on affect and vulnerability to depression. In this study we are using statins as an experimental tool to investigate this relationship further. Statins are widely prescribed agents that are regarded as very safe and so are suitable tools in this context. We have selected simvastatin because it is one of the most widely used statins and has an excellent safety profile, being also available 'over the counter'.

DETAILED DESCRIPTION:
Depression is common and associated with considerable disability (James-2018). Furthermore, the impact of the current Covid-19 pandemic on the mental health of the general population, especially in terms of depression, anxiety, and stress is proving enormous (Vindegaard-2020). Such effect is likely due to an intricate combination of biological factors (potentially neuroimmune [Troyer-2020]) as well as psychosocial aspects (such as self-isolation and loneliness [Blanco-2020]) - the latter significantly associated with worse mental health outcomes (Leigh-Hunt-2017). In particular, an important factor associated with increased vulnerability to depression is social isolation and loneliness, both of which are exacerbated by the measures needed to control the Covid-19 pandemic. Within this context, there is a need to identify factors that may be protective against the negative mental health consequences of such psychosocial stressors.

There is increasing evidence that low-level inflammation is an important mechanism by which psychosocial stress, including loneliness, predisposes to depressive symptomatology (Nersesian-2018). Consistent with this, a recent observational study conducted by our group in the context of the COVID-19 pandemic found that people who were taking a statin (which have broad anti-inflammatory properties) had a relatively increased positive bias on measures of emotional processing that are known to be associated with psychological vulnerability to depression (COSIE study, R69299/RE001). This raises the interesting possibility that reduced levels of inflammation have a protective effect within the current context of the high levels of psychosocial stress associated with the pandemic. This is consistent with a wealth of epidemiological studies showing that, at a population level, prescription of statins is associated with decreased rates of anxiety and depression (Parsaik-2014).

The aim of the current study is to extend these observational studies and experimentally test in a prospective double-blind controlled design whether reducing inflammation by administering a statin lowers vulnerability to depression in at-risk individuals, as measured by well-established cognitive biomarkers.

Patients with depression and people vulnerable to depression consistently show negative biases in emotional processing, which are believed to play a key role in the development and maintenance of clinical depressive symptoms (Roiser-2013). Overall, evidence suggests that early changes in emotional processing can serve as valid surrogate markers of antidepressant efficacy (Harmer-2017). Intriguingly, our previous study showed that patients on statins were less likely to show negative cognitive biases (COSIE study, R69299/RE001): this observation provides a potential cognitive biomarker of the ability of statins to prevent depression. We and others have also shown that induction of inflammation in healthy participants is associated with negative cognitive biases and deficits in reward learning (Cooper-2017; Miller-2017). In addition, inflammation is associated with impairment in tests of learning and memory (Gorelick-2010). This could add to the likelihood of inflammation leading to depression through compromise of problem-solving skills.

While the COSIE study suggests that statin treatment is associated with decreased negative emotional processing in an at-risk population, such observational studies are subject to confounders and require prospective controlled investigations for confirmation. In the present study therefore we propose to assess the effect of 28-days administration of statin treatment compared to placebo on emotional processing, reward learning, and working memory, in 100 healthy volunteers at-risk for depression due to loneliness in the context of the Covid-19 pandemic. We will also measure waking salivary cortisol as an index of the effect of inflammation to activate the hypothalamic-pituitary-adrenal (HPA) axis. The statin we have selected is simvastatin in view of its widespread use and safety. Our prediction is that, relative to placebo, in this at-risk group, simvastatin will lead to positive effects on emotional processing, reward learning, working memory, and will also lower waking salivary cortisol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 21-65 years
* At-risk for depression as measured by a score >6 on the UCLA 3-item Loneliness Scale
* Body Mass Index in the range of 18-30
* Willing and able to give informed consent for participation in the study
* Registered with a GP and consenting to GP being informed of participation in the study
* Currently living in the UK and sufficiently fluent English to understand and complete the tasks
* Able to access and use a computer with Internet
* Able to complete online questionnaires and tasks

Exclusion Criteria:

* Currently on any regular prescribed medications (except the contraceptive pill), unless unlikely to compromise safety or affect data quality in the opinion of the Investigator;
* History or current significant psychiatric illness (other than past [>6 months] episodes of depression or anxiety)
* Current alcohol or substance misuse disorder (< 6 months)
* History of, or current significant hepatic disease
* History of, or current significant neurological condition (e.g. epilepsy)
* History of haemorrhagic stroke or deep brain structures stroke
* Known hyperglycaemia/pre-diabetes
* Known hypersensitivity to the study drug (i.e. simvastatin) or sucrose
* Pregnant, breast feeding, women of child-bearing potential not using appropriate contraceptive measures
* Participation in a study that uses the same or similar computer tasks (apart from the N-back) as those used in the present study
* Participation in a study that involves the use of a medication within the last 3 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Facial expression recognition task (FERT) | Day 28-30 of drug/placebo administration
  Accuracy on a computer-based task of emotional processing (i.e. Facial expression recognition task [FERT]), comparing those receiving drug and placebo.
Facial expression recognition task (FERT) | Day 28-30 of drug/placebo administration
  Reaction times on a computer-based task of emotional processing (i.e. Facial expression recognition task [FERT]), comparing those receiving drug and placebo.

SECONDARY OUTCOMES:
Emotional categorisation task (ECAT) | Day 28-30 of drug/placebo administration
  Accuracy on a computer-based task of emotional processing (i.e. Emotional categorisation task [ECAT]), comparing those receiving drug and placebo.
Emotional categorisation task (ECAT) | Day 28-30 of drug/placebo administration
  Reaction times on a computer-based task of emotional processing (i.e. Emotional categorisation task [ECAT]), comparing those receiving drug and placebo.
Emotional recall task (EREC) | Day 28-30 of drug/placebo administration
  Accuracy on a computer-based task of emotional processing (i.e. Emotional recall task [EREC]), comparing those receiving drug and placebo.
Emotional recall task (EREC) | Day 28-30 of drug/placebo administration
  Reaction times on a computer-based task of emotional processing (i.e. Emotional recall task [EREC]), comparing those receiving drug and placebo.
Probabilistic instrumental learning task (PILT) | Day 28-30 of drug/placebo administration
  Amount won/loss on computer-based tasks of reward learning (Probabilistic instrumental learning task [PILT]) comparing those receiving drug and placebo.
Probabilistic instrumental learning task (PILT) | Day 28-30 of drug/placebo administration
  Number of choice switches on computer-based tasks of reward learning (Probabilistic instrumental learning task [PILT]) comparing those receiving drug and placebo.
N-back | Day 28-30 of drug/placebo administration
  Accuracy on computer-based tasks of working memory (N-back) comparing those receiving drug and placebo.
N-back | Day 28-30 of drug/placebo administration
  Reaction times on computer-based tasks of working memory (N-back) comparing those receiving drug and placebo.
Salivary cortisol | Day 28-30 of drug/placebo administration
  Changes in salivary cortisol from baseline to 28-30 days, comparing those receiving drug and placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised research data without any personal data (e.g., reaction time data) will also be stored on private Open Science Framework (OSF) project components that are accessible only to the research team. Parts of the data might be uploaded to online data repositories or made publicly available on OSF in a completely anonymised fashion, to facilitate open science. Data uploaded in this way will be stored on OSF indefinitely.